CLINICAL TRIAL: NCT06967571
Title: Reconstruction With a Lawrence-Hunt Jejunal Pouch for Upfront Total Gastrectomy - Study Protocol of a Prospective, Single-arm, Phase II Trial
Brief Title: Reconstruction With a Lawrence-Hunt Jejunal Pouch After Total Gastrectomy
Acronym: REJOY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7445
Record Dates: First submitted 2025-03-19; First posted 2025-05-13 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-03

CONDITIONS: Total Gastrectomy; Gastric Cancer
Keywords: gastric cancer; total gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open or laparoscopic TG followed by JP reconstruction. (Experimental): All participants will undergo open or laparoscopic Total Gastrectomy (TG) followed by Jejunal Pouch (JP) reconstruction.
  Interventions: Procedure: Jejunal Pouch reconstruction.

INTERVENTIONS:
Procedure: Jejunal Pouch reconstruction. — The JP will be fashioned with a standard length of 12 cm using two 60 mm staple lines, the esophago-pouch anastomosis will be performed with a circular mechanical 25 mm stapling device, and finally the staple entrance on the pouch will be closed with two layers of running sutures in Vicryl 3/0

SUMMARY:
The aim of the study is to establish the efficacy of jejunal pouch reconstruction in reducing dumping syndrome in patients undergoing total gastrectomy, ultimately enhancing postoperative quality of life and nutritional status.

DETAILED DESCRIPTION:
Total gastrectomy (TG) with Roux-en-Y (RY) esophageal-jejunal anastomosis is performed for various gastric malignancies or as a prophylactic strategy in patients with hereditary diffuse gastric cancer syndrome harboring CDH1 mutation at risk of developing gastric cancer. The surgical procedure is, however, complicated in the post-operative months by weight loss and nutritional deficiency in most patients, requiring frequent follow-up, and by functional issues such as reflux and dumping syndrome in about 30% of cases, which significantly impact the patient's quality of life. To prevent the poorer outcomes reported by patients undergoing total gastrectomy, one strategy could be a modification of the reconstruction method using a jejunal pouch reconstruction (JP) that may mitigate symptoms by slowing gastric emptying and enhancing nutrient absorption. JP has so far proven several benefits in improving postoperative outcomes (reflux and dumping syndrome), nutritional outcomes, and QoL up to 2 years after surgery. The technique has been mostly studied in the Eastern countries (Japan and South Korea) and, since 2021, has been recommended by the French Association of Surgery as the technique of choice for reconstruction after total gastrectomy. However, in most European centers, this technique has not yet been introduced as a routine procedure due to a relative lack of data on the clinical benefit and risk profile in the Western population.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years.
* Histologically confirmed gastric tumor (including adenocarcinoma, gastrointestinal stromal tumor - GIST- or neuroendocrine tumor) or patients with CDH1 mutation, scheduled for TG with a maximal esophageal resection of < 6 cm.
* Informed consent capability.

Exclusion Criteria:

* Prior abdominal surgeries affecting the jejunum.
* Severe comorbidities or non-appropriate organ function: uncontrolled diabetes with HbA1C > 7.5, significant heart disease: New York Heart Association (NYHA) functional classification Class III or IV, chronic obstructive pulmonary disease (COPD) requiring oxygen supplementation or continuous positive airway pressure (CPAP), chronic corticosteroid therapy (daily for more than 6 months), neutrophil count < 2000/mm3, hemoglobin < 8.0 g/dL, platelet count < 100,000/mm3, serum total bilirubin > 1.5 mg/dL, serum aspartate aminotransferase (AST) >100 IU/L, serum alanine aminotransferase (ALT) >100 IU/L, and creatinine clearance (CCr) ≥ 50 mL/min), ECOG performance status > 1.
* Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Dumping syndrome reduction rate | 12 months after surgery
  Evaluate the reduction in the incidence of dumping syndrome after TG with JP reconstruction with the Sigstad questionnaire.

SECONDARY OUTCOMES:
Dumping syndrome severity | The DSS was administered at 3, 6, and 12 months after surgery.
  Dumping syndrome severity was assessed using the Arts Dumping Severity Score (DSS), an 11-item questionnaire with a total score range of 0-33, where higher scores indicate worse symptoms.
Nutritional status - weight | 3, 6 & 12 months after surgery
  Assess the nutritional status using weight in kilograms
Nutritional status - height | 3, 6 & 12 months after surgery
  Assess the nutritional status using height in meters
Nutritional status - Body Mass Index (BMI) | 3, 6 & 12 months after surgery
  To Assess the nutritional status weight and height will be combined to report BMI in kg/m^2
Nutritional status | 3, 6 & 12 months after surgery
  Assess the nutritional status using validated metrics such as the serum iron levels, albumin levels, B12 levels and vitamin D levels.
Gastrointestinal Quality of Life Index (GIQLI) | 3, 6 & 12 months after surgery
  Evaluate the quality of life using using the Italian versions of the GIQLI questionnaire. The maximum GIQLI in the international score is 144 and its worst value is 0.
EORTC QLQ-C30 | Assessments were performed at 3, 6, and 12 months after surgery
  Quality of life was assessed using the Italian version of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30). All scales were transformed into scores ranging from 0 to 100. For the functional scales and the global health status/quality of life scale, higher scores indicate a better outcome, whereas for the symptom scales higher scores indicate greater symptom severity.
Postoperative complications | 12 months after surgery
  Measure the rate of postoperative complications. All severe adverse events (SAEs) will be collected starting with the surgical admission until the end of the study period (12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Agnes, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trapani R, Rausei S, Reddavid R, Degiuli M; ITALIAN RESEARCH GROUP FOR GASTRIC CANCER (GIRCG) Clinical Investigators. Risk factors for esophago-jejunal anastomosis leakage after total gastrectomy for cancer. A multicenter retrospective study of the Italian research group for gastric cancer. Eur J Surg Oncol. 2020 Dec;46(12):2243-2247. doi: 10.1016/j.ejso.2020.06.035. Epub 2020 Jul 9. PMID 32703713
- [Result] A'Hern RP. Sample size tables for exact single-stage phase II designs. Stat Med. 2001 Mar 30;20(6):859-66. doi: 10.1002/sim.721. PMID 11252008
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Apolone G, Filiberti A, Cifani S, Ruggiata R, Mosconi P. Evaluation of the EORTC QLQ-C30 questionnaire: a comparison with SF-36 Health Survey in a cohort of Italian long-survival cancer patients. Ann Oncol. 1998 May;9(5):549-57. doi: 10.1023/a:1008264412398. PMID 9653497
- [Result] Ponticelli C, Colombo D, Novara M, Basilisco G; CETRA Study Group. Gastrointestinal symptoms impair quality of life in Italian renal transplant recipients but are under-recognized by physicians. Transpl Int. 2010 Nov;23(11):1126-34. doi: 10.1111/j.1432-2277.2010.01115.x. Epub 2010 Aug 19. PMID 20525020
- [Result] Scarpellini E, Arts J, Karamanolis G, Laurenius A, Siquini W, Suzuki H, Ukleja A, Van Beek A, Vanuytsel T, Bor S, Ceppa E, Di Lorenzo C, Emous M, Hammer H, Hellstrom P, Laville M, Lundell L, Masclee A, Ritz P, Tack J. International consensus on the diagnosis and management of dumping syndrome. Nat Rev Endocrinol. 2020 Aug;16(8):448-466. doi: 10.1038/s41574-020-0357-5. Epub 2020 May 26. PMID 32457534
- [Result] Sigstad H. A clinical diagnostic index in the diagnosis of the dumping syndrome. Changes in plasma volume and blood sugar after a test meal. Acta Med Scand. 1970 Dec;188(6):479-86. No abstract available. PMID 5507449
- [Result] Voron T, Romain B, Bergeat D, Veziant J, Gagniere J, Le Roy B, Pasquer A, Eveno C, Gaujoux S, Pezet D, Gronnier C; sous l'egide de l'Association francaise de chirurgie (AFC); Collaborateurs (relecteurs). Surgical management of gastric adenocarcinoma. Official expert recommendations delivered under the aegis of the French Association of Surgery (AFC). J Visc Surg. 2020 Apr;157(2):117-126. doi: 10.1016/j.jviscsurg.2020.02.006. Epub 2020 Mar 6. PMID 32151595
- [Result] Syn NL, Wee I, Shabbir A, Kim G, So JB. Pouch Versus No Pouch Following Total Gastrectomy: Meta-analysis of Randomized and Non-randomized Studies. Ann Surg. 2019 Jun;269(6):1041-1053. doi: 10.1097/SLA.0000000000003082. PMID 31082900
- [Result] Tanizawa Y, Tanabe K, Kawahira H, Fujita J, Takiguchi N, Takahashi M, Ito Y, Mitsumori N, Namikawa T, Oshio A, Nakada K; Japan Postgastrectomy Syndrome Working Party. Specific Features of Dumping Syndrome after Various Types of Gastrectomy as Assessed by a Newly Developed Integrated Questionnaire, the PGSAS-45. Dig Surg. 2016;33(2):94-103. doi: 10.1159/000442217. Epub 2015 Dec 18. PMID 26682541